CLINICAL TRIAL: NCT03561792
Title: Diaphragmatic Rapid Shallow Breathing Index for Predicting Weaning Outcome From Mechanical Ventilation: Comparison With Traditional Rapid Shallow Breathing Index
Brief Title: Diaphragmatic Rapid Shallow Breathing Index for Predicting Weaning Outcome From Mechanical Ventilation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zagazig University (Other Government)
Responsible Party: Principal Investigator, Sherif M. S. Mowafy, Lecturer of Anesthesia and Surgical Intensive Care, Zagazig University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 4664/28-5-2018
Record Dates: First submitted 2018-06-05; First posted 2018-06-19 (Actual); Last update posted 2019-01-02 (Actual); Status verified 2018-12

CONDITIONS: Weaning Failure

STUDY DESIGN:
Who Masked: Care Provider
Masking Description: The ICU team on charge takes the decision to continue spontaneous breathing trial (SBT) according to the local practice protocols which depends on the traditional RSBI (RSBI < 105 predicts successful weaning). The ICU team will not be allowed to know the results of diaphragmatic ultrasound.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- traditional RSBI (No Intervention): the decision to continue SBT depends on the traditional RSBI (RSBI < 105 predicts successful weaning)
- Diaphragmatic RSBI (Experimental): diaphragm ultrasound was done to measure diaphragmatic displacement which is used to calculate DRSBI and The investigator takes the decision about SBT continuation based on the result of DRSBI (DRSBI < 1.3 predicts successful weaning)
  Interventions: Other: Diaphragm ultrasound

INTERVENTIONS:
Other: Diaphragm ultrasound — In the semi-sitting position ultrasonography for diaphragmatic displacement was performed by the same intensivist. Diaphragmatic movement was evaluated by using 2 to 5 MHz US probe (Sonosite M-Turbo machine). The right hemidiaphragm was examined by two-dimensional (2D) and M-mode to record diaphragm displacement.in M-mode, the diaphragmatic displacement (cm) was measured and then DRSBI was calculated by respiratory rate (RR)/ diaphragmatic displacement (DD) (in mm)
  Arms: Diaphragmatic RSBI

SUMMARY:
Predicting successful discontinuation from mechanical ventilation has been a focus of interest to all critical care physicians . Various weaning indices have been investigated to optimize the weaning process. Among them, the rapid shallow breathing index (RSBI) has gained wide use but it have different sensitivities and specificities. By substituting tidal volume (VT) with diaphragmatic displacement (DD) in the calculation of RSBI a new index (the diaphragmatic rapid shallow breathing index DRSBI) was proposed and it was independently associated with weaning failure and its accuracy for predicting weaning outcome is expected to be superior to the traditional RSBI.

DETAILED DESCRIPTION:
The rapid shallow breathing index (RSBI), calculated from respiratory rate divided by tidal volume (RR/VT), is a well-known weaning index and one of the most clinical indices used to predict weaning outcome. However, it has some limitations in predicting weaning outcomes. Several previous studies have defined different sensitivities and specificities for RSBI less than 105 to predict weaning success which may lead to errors in predicting successful weaning.

On the other hand, Weaning failure is likely to occur if there is an imbalance between the load on the inspiratory muscles and their neuromuscular capacity, the imbalance between the mechanical load imposed on the diaphragm which is the major muscle of inspiration and its ability to cope with it. Therefore, evaluating the function of diaphragm before any weaning trial could be useful in predicting weaning outcome.

Bedside ultrasonography is an easy, fast, noninvasive, and accurate maneuver for evaluating diaphragmatic function. Diaphragmatic displacement (DD) reflecting the ability of diaphragm to produce force and subsequently tidal volume during inspiration and defined as displacement of less than 10 mm has been found to be a predictor of weaning failure among patients in medical ICUs.

Spadaro et al. proposed substituting VT with DD in the RSBI, and calculating diaphragmatic RSBI (DRSBI) would result in a more accurate predictive index than the traditional RSBI.

ELIGIBILITY:
Inclusion Criteria:

* Patient or relative acceptance
* Mechanically ventilated for more than 48 hours
* Ready to wean and at their first spontaneous breathing trial
* meeting all weaning criteria

Exclusion Criteria:

* history of any neuromuscular disease
* diaphragmatic palsy
* cervical injury
* current chest trauma
* thoracotomy for any reason
* patients in whom neuromuscular blockers are used in the last 48 hours before the study
* patients for whom aminoglycosides are prescribed during their course in ICU

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 106 (Actual)
Dates: Start 2017-12-01 (Actual); Primary Completion 2018-08-30 (Actual); Study Completion 2018-10-01 (Actual)

PRIMARY OUTCOMES:
weaning failure | 48 hours
  weaning failure is the inability to maintain spontaneous breathing for at least 48 h, Patients who required reintubation or noninvasive positive pressure ventilation within 48 h of discontinuation of mechanical ventilation (MV) will be considered failed to wean

CONTACTS AND LOCATIONS:
Overall Officials: Essam F Abdelgalel, MD, Study Director — Anesthesia and Surgical Intensive Care Department, faculty of medicine, Zagazig University; Sherif MS Mowafy, MD, Principal Investigator — Anesthesia and Surgical Intensive Care Department, faculty of medicine, Zagazig University
Locations (1):
- Zagazig University Hospitals, Zagazig, Sharqia Province, Egypt

IPD SHARING:
Plan to Share IPD: Yes
all collected IPD
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: starting 6 months after publication
Access Criteria: from the study director

REFERENCES:
- [Background] Kulkarni AP, Agarwal V. Extubation failure in intensive care unit: predictors and management. Indian J Crit Care Med. 2008 Jan;12(1):1-9. doi: 10.4103/0972-5229.40942. PMID 19826583
- [Background] Penuelas O, Frutos-Vivar F, Fernandez C, Anzueto A, Epstein SK, Apezteguia C, Gonzalez M, Nin N, Raymondos K, Tomicic V, Desmery P, Arabi Y, Pelosi P, Kuiper M, Jibaja M, Matamis D, Ferguson ND, Esteban A; Ventila Group. Characteristics and outcomes of ventilated patients according to time to liberation from mechanical ventilation. Am J Respir Crit Care Med. 2011 Aug 15;184(4):430-7. doi: 10.1164/rccm.201011-1887OC. PMID 21616997
- [Background] Thille AW, Harrois A, Schortgen F, Brun-Buisson C, Brochard L. Outcomes of extubation failure in medical intensive care unit patients. Crit Care Med. 2011 Dec;39(12):2612-8. doi: 10.1097/CCM.0b013e3182282a5a. PMID 21765357
- [Background] McConville JF, Kress JP. Weaning patients from the ventilator. N Engl J Med. 2012 Dec 6;367(23):2233-9. doi: 10.1056/NEJMra1203367. No abstract available. PMID 23215559
- [Background] Spadaro S, Grasso S, Mauri T, Dalla Corte F, Alvisi V, Ragazzi R, Cricca V, Biondi G, Di Mussi R, Marangoni E, Volta CA. Can diaphragmatic ultrasonography performed during the T-tube trial predict weaning failure? The role of diaphragmatic rapid shallow breathing index. Crit Care. 2016 Sep 28;20(1):305. doi: 10.1186/s13054-016-1479-y. PMID 27677861
- [Background] Yang KL, Tobin MJ. A prospective study of indexes predicting the outcome of trials of weaning from mechanical ventilation. N Engl J Med. 1991 May 23;324(21):1445-50. doi: 10.1056/NEJM199105233242101. PMID 2023603
- [Background] Lee KH, Hui KP, Chan TB, Tan WC, Lim TK. Rapid shallow breathing (frequency-tidal volume ratio) did not predict extubation outcome. Chest. 1994 Feb;105(2):540-3. doi: 10.1378/chest.105.2.540. PMID 8306759
- [Background] Pirompanich P, Romsaiyut S. Correction to: Use of diaphragm thickening fraction combined with rapid shallow breathing index for predicting success of weaning from mechanical ventilator in medical patients. J Intensive Care. 2018 Apr 23;6:25. doi: 10.1186/s40560-018-0293-9. eCollection 2018. PMID 29714351
- [Background] Zambon M, Greco M, Bocchino S, Cabrini L, Beccaria PF, Zangrillo A. Assessment of diaphragmatic dysfunction in the critically ill patient with ultrasound: a systematic review. Intensive Care Med. 2017 Jan;43(1):29-38. doi: 10.1007/s00134-016-4524-z. Epub 2016 Sep 12. PMID 27620292
- [Background] Kim WY, Suh HJ, Hong SB, Koh Y, Lim CM. Diaphragm dysfunction assessed by ultrasonography: influence on weaning from mechanical ventilation. Crit Care Med. 2011 Dec;39(12):2627-30. doi: 10.1097/CCM.0b013e3182266408. PMID 21705883
- [Background] Yoo JW, Lee SJ, Lee JD, Kim HC. Comparison of clinical utility between diaphragm excursion and thickening change using ultrasonography to predict extubation success. Korean J Intern Med. 2018 Mar;33(2):331-339. doi: 10.3904/kjim.2016.152. Epub 2017 Oct 19. PMID 29050461
- [Background] Boles JM, Bion J, Connors A, Herridge M, Marsh B, Melot C, Pearl R, Silverman H, Stanchina M, Vieillard-Baron A, Welte T. Weaning from mechanical ventilation. Eur Respir J. 2007 May;29(5):1033-56. doi: 10.1183/09031936.00010206. PMID 17470624
- [Background] MacIntyre NR, Cook DJ, Ely EW Jr, Epstein SK, Fink JB, Heffner JE, Hess D, Hubmayer RD, Scheinhorn DJ; American College of Chest Physicians; American Association for Respiratory Care; American College of Critical Care Medicine. Evidence-based guidelines for weaning and discontinuing ventilatory support: a collective task force facilitated by the American College of Chest Physicians; the American Association for Respiratory Care; and the American College of Critical Care Medicine. Chest. 2001 Dec;120(6 Suppl):375S-95S. doi: 10.1378/chest.120.6_suppl.375s. No abstract available. PMID 11742959
- [Background] Boussuges A, Gole Y, Blanc P. Diaphragmatic motion studied by m-mode ultrasonography: methods, reproducibility, and normal values. Chest. 2009 Feb;135(2):391-400. doi: 10.1378/chest.08-1541. Epub 2008 Nov 18. PMID 19017880
- [Background] Matamis D, Soilemezi E, Tsagourias M, Akoumianaki E, Dimassi S, Boroli F, Richard JC, Brochard L. Sonographic evaluation of the diaphragm in critically ill patients. Technique and clinical applications. Intensive Care Med. 2013 May;39(5):801-10. doi: 10.1007/s00134-013-2823-1. Epub 2013 Jan 24. PMID 23344830